CLINICAL TRIAL: NCT00436904
Title: Antibody Therapy With Alemtuzumab and Rituximab for Initial Treatment of High Risk Chronic Lymphocytic Leukemia
Brief Title: Alemtuzumab and Rituximab in Treating Patients With High-Risk, Early-Stage Chronic Lymphocytic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000529809; P30CA015083 (NIH); MC038G (Other: Mayo Clinic Cancer Center); 801-04 (Other: Mayo Clinic IRB); 106.G0309 (Other: Bayer and Berlex protocol); U3023s (Other: Genentech Protocol)
Record Dates: First submitted 2007-02-15; First posted 2007-02-19 (Estimated); Results first posted 2011-10-26 (Estimated); Last update posted 2011-12-01 (Estimated); Status verified 2011-11

CONDITIONS: Leukemia
Keywords: stage 0 chronic lymphocytic leukemia; stage I chronic lymphocytic leukemia; stage II chronic lymphocytic leukemia; B-cell chronic lymphocytic leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Alemtuzumab; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Alemtuzumab + Rituximab (Experimental): Alemtuzumab 30mg Monday, Wednesday, and Friday x 5 weeks, Rituximab 375/mg/m2 IV weekly (Wednesday) x 4 weeks (weeks 2-5)
  Interventions: Drug: Alemtuzumab; Drug: Rituximab

INTERVENTIONS:
Drug: Alemtuzumab — 30 mg Monday, Wednesday, and Friday x 5 weeks
Drug: Rituximab — 375mg/m2 IV weekly (Wednesday) x 4 weeks (weeks 2-5)

SUMMARY:
RATIONALE: Monoclonal antibodies, such as alemtuzumab and rituximab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. Giving alemtuzumab together with rituximab may kill more cancer cells.

PURPOSE: This phase II trial is studying the side effects and how well giving alemtuzumab together with rituximab works in treating patients with high-risk, early-stage chronic lymphocytic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the rate of complete and overall response to alemtuzumab and rituximab in patients with high-risk, early-stage chronic lymphocytic leukemia.
* Determine the toxicity of this regimen in these patients. Secondary
* Determine the overall survival and time to progression of patients treated with this regimen.
* Determine time to response and duration of response in patients treated with this regimen.
* Correlate prognostic markers 11q-, 17p-, unmutated VH gene, and CD38+ with clinical outcome.
* Determine response to this regimen using an expanded definition of response that includes minimal residual disease detected by sensitive flow cytometry in patients in complete clinical remission and single rearranged IgVH gene detected by polymerase chain reaction in patients with no monoclonal population on flow cytometry.
* Correlate in vitro response with clinical outcome in patients treated with this regimen.
* Determine if alemtuzumab and rituximab are synergistic in vitro.
* Determine the mechanism of action of this regimen in vitro.
* Determine the effect of this regimen on immune function.
* Monitor T-lymphocyte, natural killer cell, and monocyte number during and after treatment in these patients.
* Serially evaluate T-lymphocyte immunophenotype and function in patients treated with this regimen.
* Monitor recovery of humoral immunity by serial serum protein electrophoresis, immunofixation electrophoresis, and immunoglobulin quantification.

OUTLINE:

* Dose-escalation (week 1): Patients receive rituximab IV on day 1 and escalating doses of alemtuzumab subcutaneously (SC) on days 3-5 in week 1.
* Treatment (weeks 2-5): Patients receive alemtuzumab SC on days 1-3 (at the highest dose administered during week 1) and rituximab IV on day 3 in weeks 2-5 in the absence of disease progression or unacceptable toxicity.

Patients undergo blood collection at baseline and periodically during study treatment for pharmacokinetic and prognostic biomarker (11q-, 17p-, unmutated IgVH, and CD38 expression by flow cytometry and fluorescent in-situ hybridization) studies. Immune function (CDR3 T-cell receptor by reverse transcriptase-polymerase chain reaction) and in vitro and in vivo response are also examined.

After completion of study therapy, patients are followed periodically for 5 years.

PROJECTED ACCRUAL: A total of 33 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of B-cell chronic lymphocytic leukemia (CLL)

- Early-stage, biologically high-risk disease defined by the following criteria:

* Rai stage 0-II (does not meet standard NCI-sponsored Working Group criteria for treatment)
* Clinical and phenotypic features manifested in the peripheral blood, including the following:

  * Minimum threshold peripheral blood lymphocyte count of > 5,000/mm³
  * Small-to-moderate peripheral blood lymphocytes with ≤ 55% prolymphocytes
  * Monoclonality of B lymphocytes by immunophenotypic evaluation, demonstrating co-expression of CD19, CD5, and CD23 antigens, surface expression of CD20 and CD52, and B-cell monoclonal population defined by light-chain exclusions
* Poor prognosis demonstrated by ≥ 1 of the following high-risk parameters:

  * Unmutated human immunoglobulin variable region heavy chain (IgVH) gene and CD38 expression (≥ 30% cells positive on flow cytometry) OR unmutated IgVH ZAP-70 expression (≥ 20% cells positive on flow cytometry) = 11q- = 17p-

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Creatinine ≤ 1.5 times upper limit of normal (ULN)
* Total bilirubin ≤ 3.0 times ULN OR direct bilirubin ≤ 1.5 times ULN
* AST ≤ 3.0 times ULN (unless due to hemolysis or CLL)
* Hemoglobin ≥ 9.0 g/dL
* No New York Heart Association class III-IV heart disease
* No myocardial infarction within the past month
* No uncontrolled infection
* No active HIV infection
* No evidence of autoimmune hemolytic anemia, immune thrombocytopenia, or pure red blood cell aplasia
* No other active primary malignancy requiring treatment or limiting survival to less than 2 years

PRIOR CONCURRENT THERAPY:

* No prior treatment for CLL
* Prior corticosteroids allowed
* No prior radiotherapy
* More than 4 weeks since prior major surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2004-12; Primary Completion 2008-07 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clive S. Zent, MD, Study Chair — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Result] Zent CS, Call TG, Shanafelt TD, Tschumper RC, Jelinek DF, Bowen DA, Secreto CR, Laplant BR, Kabat BF, Kay NE. Early treatment of high-risk chronic lymphocytic leukemia with alemtuzumab and rituximab. Cancer. 2008 Oct 15;113(8):2110-8. doi: 10.1002/cncr.23824. PMID 18759253
- [Result] Zent CS, Secreto CR, LaPlant BR, Bone ND, Call TG, Shanafelt TD, Jelinek DF, Tschumper RC, Kay NE. Direct and complement dependent cytotoxicity in CLL cells from patients with high-risk early-intermediate stage chronic lymphocytic leukemia (CLL) treated with alemtuzumab and rituximab. Leuk Res. 2008 Dec;32(12):1849-56. doi: 10.1016/j.leukres.2008.05.014. Epub 2008 Jun 27. PMID 18584865

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Alemtuzumab + Rituximab
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Alemtuzumab + Rituximab
Number analyzed (Participants) | 30
Age Continuous [Median (Full Range); unit: years] | 61 [29 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 20
Region of Enrollment [Number; unit: participants]
  United States | 30
Performance Score [Number; unit: participants] — Classifies patients according to their functional impairment. Scores range from 0 (fully active) to 5 (death).
  participants
    0 - Fully Active | 27
    1 - Ambulatory, restricted strenuous activity | 3

OUTCOME MEASURES:

1. Primary Outcome: Confirmed Response, Defined as Objective Complete Remission or Partial Remission for a Duration of at Least 2 Months
Description: Confirmed response is defined as a > 50% decrease in clinical symptoms from baseline and recovery from blood counts.
Time Frame: Up to 6 months
Population: Number of patients with a confirmed response out of total patients evaluable for response.
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | Alemtuzumab + Rituximab
Number analyzed (Participants) | 30
participants | 27 [23.1 to 29.1]

2. Primary Outcome: Number of Participants With Treatment Related Adverse Events
Description: Adverse events (AE) that are classified as either possibly, probably, or definitely related to study treatment according to the National Cancer Institute Common Toxicity Criteria for Adverse Events (NCI CTCAE version 3.0). The maximum grade for each type of AE will be recorded for each patient. Grade refers to the severity of the AE.>
  > Grade 1: Mild AE, Grade 2: Moderate AE, Grade 3: Severe AE, Grade 4: Life-threatening or disabling AE, Grade 5: Death related AE
Time Frame: Weekly for first 6 weeks, then monthly for 6 months, then at 9 and 12 months post registration
Measure: Number; unit: participants
Arm/Group | Alemtuzumab + Rituximab
Number analyzed (Participants) | 30
participants
  Grade 3-4 Hematologic | 11
  Grade 3-4 Non-hematologic | 3

3. Secondary Outcome: Time to Response
Description: Calculated from the date of registration until the first date at which the patient's objective status was classified as a response. In patients who do not achieve a response, time to response will be censored at the patient's last evaluation date. Response is defined the same way as in the response primary outcome measure.
Time Frame: Registration to first response (up to 5 years)
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Alemtuzumab + Rituximab
Number analyzed (Participants) | 30
Days | 8 [8 to 14]

4. Secondary Outcome: Duration of Response
Description: Duration of response is calculated from the date of documented response until the date of progression in the subset of patients who respond to treatment. In patients who have not yet progressed, duration of response will be censored at the patient's last evaluation date.
Time Frame: Up to 5 years
Population: Patients that responded were included in the analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Alemtuzumab + Rituximab
Number analyzed (Participants) | 27
Months | 14.4 [9.3 to 22.5]

5. Secondary Outcome: Survival
Description: Survival is calculated from the date of registration to the date of death due to any cause. In patients who are still alive, survival will be censored at the last date when the patient was known to be alive.
Time Frame: Death or last follow-up (up to 5 years)
Population: At analysis time, only 1 out of 30 patients had died. Thus, median survival was not attainable.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Alemtuzumab + Rituximab
Number analyzed (Participants) | 0

6. Secondary Outcome: Time to Disease Progression
Description: Calculated from date of registration to date of disease progression. In patients that have not progressed, time to disease progression will be censored at the patient's last evaluation date.
Time Frame: Time from registration to progression (up to 5 years)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Alemtuzumab + Rituximab
Number analyzed (Participants) | 30
Months | 12.5 [7.2 to 19.3]

ADVERSE EVENTS:
Arm/Group | Alemtuzumab + Rituximab
Serious Adverse Events (participants affected / at risk) | 1/30
Other Adverse Events (participants affected / at risk) | 29/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alemtuzumab + Rituximab (N=30)
Skin infection (Infections and infestations) | 1 (1)
Ischemia-Cerebral (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alemtuzumab + Rituximab (N=30)
Anemia (Blood and lymphatic system disorders) | 3 (4)
Diarrhea-No Colostom (Gastrointestinal disorders) | 6 (8)
Dyspepsia (Gastrointestinal disorders) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Pain-Abdominal (Gastrointestinal disorders) | 3 (3)
Vomiting (Gastrointestinal disorders) | 1 (1)
Fever-No ANC (General disorders) | 15 (24)
Rigors (General disorders) | 1 (1)
Hypersensitivity (Immune system disorders) | 3 (3)
Blood Infection (Infections and infestations) | 2 (2)
Bronchial infection (Infections and infestations) | 2 (2)
Bronchus infection (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 3 (4)
Respiratory tract infection (Infections and infestations) | 6 (6)
Skin infection (Infections and infestations) | 4 (5)
Upper airway infection (Infections and infestations) | 1 (1)
Appendix injury (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (3)
Aspartate aminotransferase increased (Investigations) | 2 (2)
Blood bilirubin increased (Investigations) | 3 (4)
Leukopenia (Investigations) | 19 (55)
Lymphopenia (Investigations) | 1 (1)
Neutropenia (Investigations) | 12 (24)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 (1)
Olfactory nerve disorder (Nervous system disorders) | 1 (1)
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash/Desquamation (Skin and subcutaneous tissue disorders) | 24 (57)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes